CLINICAL TRIAL: NCT01304303
Title: Pharmacokinetic and Safety Study of SPARC1023 Alone and in Carboplatin Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLR_10_23
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor in Advanced Stage
Keywords: solid; tumor; taxane; platinum
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPARC1023 I (Experimental)
  Interventions: Drug: SPARC1023 I
- SPARC1023 II (Experimental)
  Interventions: Drug: SPARC1023 II

INTERVENTIONS:
Drug: SPARC1023 I — IV administration
  Arms: SPARC1023 I
Drug: SPARC1023 II — IV administration
  Arms: SPARC1023 II

SUMMARY:
Phase I study of SPARC1023 alone and in combination with carboplatin

DETAILED DESCRIPTION:
Pharmacokinetic profile and dose escalation study of SPARC1023 when administered as 30-min infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ECOG Performance Status ≤ 1.
* Estimated life expectancy of at least 12-weeks;
* Measurable disease as per RECIST guideline (Version 1.1);

Exclusion Criteria:

* Any malignancy within past 5-years, except non-melanoma skin cancer, cervical intraepithelial neoplasia, or in situ cervical cancer
* Known hypersensitivity to the study drugs
* Treatment with any anti-cancer agents within 28 days of study entry
* Presence of clinically evident active CNS metastases, including leptomeningeal involvement, requiring steroid or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Determination of MTD | One 21-day treatment cycle
  MTD for SPARC1023 in combination with carboplatin will be determined. MTD will be defined as the SPARC1023 dose below the dose at which DLT (Dose Limiting Toxicity) is seen for ≥ 2 subjects.

SECONDARY OUTCOMES:
Establishing the pharmacokinetic profile | One 21-day treatment cycle
  Plasma levels of SPARC1023 and Carboplatin will be determined and PK parameters viz. Cmax, AUC0-t, AUC 0-∞, MRT, Tmax, t½ , Kel, Vd for SPARC1023 in combination with carboplatin will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC Site 1, Buffalo, New York, United States